CLINICAL TRIAL: NCT01674881
Title: A Randomized Controlled Trial of Mindfulness-based Cognitive Therapy (MBCT) on Chronic Pain in Women Treated for Breast Cancer
Brief Title: The Effectiveness of Mindfulness on Chronic Pain in Breast Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EPoS-1
Record Dates: First submitted 2012-08-24; First posted 2012-08-29 (Estimated); Last update posted 2015-04-14 (Estimated); Status verified 2013-08

CONDITIONS: Breast Cancer; Chronic Pain
Keywords: Mindfulness; breast cancer; chronic pain; mediators; distress; Breast cancer survivors; Effectiveness of MBCT on chronic pain; Potential mediators and moderators; Effectiveness of MBCT on psychological symptoms
MeSH Terms: conditions — Breast Neoplasms; Chronic Pain | interventions — Mindfulness-Based Cognitive Therapy; Waiting Lists

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mindfulness-Based Cognitive Therapy (MBCT) (Experimental): This group will receive MBCT for 8 consecutive weeks.
  Interventions: Other: Mindfulness-Based Cognitive Therapy
- Waitlist control group (Other): This group is a waitlist control group.
  Interventions: Other: Waitlist

INTERVENTIONS:
Other: Mindfulness-Based Cognitive Therapy — MBCT consists of 8 sessions, incl. 1 whole-day session, weekly meetings of app. 2 hours duration. Daily homework (app. 30-45 min).
  Group format (app. 20 persons pr. group). Two trained instructors will manage the groups, both are MSc cand.psych, PhD.
  Arms: Mindfulness-Based Cognitive Therapy (MBCT)
Other: Waitlist — Waitlist: participants are offered the intervention (MBCT) after the completion of the main study
  Arms: Waitlist control group

SUMMARY:
A recent epidemiologic survey has indicated that approx. 42% of Danish women treated for breast cancer experience negative sequelae in the form of pain following treatment. Chronic pain is known to be associated with impaired social and emotional functioning, and thus presents a particular concern.

Mindfulness-based intervention is among the complementary, psychological treatments, which cancer patients commonly seek out in relation to the course of their illness. Despite the popularity of mindfulness-based intervention among cancer patients, no studies have so far investigated the effect of mindfulness-based intervention on chronic pain in breast cancer patients. While no studies so far have focused on pain, there is evidence to suggest that mindfulness-based intervention is associated with improved psychosocial adaption to cancer. Furthermore, non-cancer research suggests that mindfulness-based intervention is associated with reduced pain experiences.

The aim of this project is to investigate the effect of Mindfulness-Based Cognitive Therapy (MBCT) on chronic pain in breast cancer patients. Women who have completed their treatment for breast cancer and who experience chronic pain, will be randomized to an intervention group (MBCT) or a treatment-as-usual control group. All participants will be assessed at the same time points, i.e. before the intervention (baseline), and three times after the intervention/control condition, with the last follow-up 6 months after the intervention. In addition, a number of potential moderators and mediators of the outcome will be explored. For example, recent studies indicate that adult attachment style may constitute an important moderator and/or mediator in the development of pain, and preliminary research has suggested that attachment style may moderate the effect of mindfulness-based intervention.

The results will provide valuable new knowledge about the potential of MBCT as a treatment strategy for chronic pain in breast cancer patients, will contribute to the clarification of underlying mechanisms in the experience of and coping with pain, which could help the development of more effective, individualized interventions.

ELIGIBILITY:
Inclusion Criteria:

* A timeframe of >3 months from surgery, radiation- and chemotherapy and a minimum score of >3 on a pain scale from 0-10 corresponding to moderate pain

Exclusion Criteria:

* Breast cancer recurrence, bilateral breast cancer, other cancer, psychiatric illnesses, insufficient ability to speak and understand Danish, and chronic pain otherwise associated with the musculoskeletal system

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2012-09; Primary Completion 2014-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Pain | From baseline until 6 months
  Revised McGill Pain Questionnaire Short Form
  VAS: pain interference
  Additional items: Pain descriptors

SECONDARY OUTCOMES:
Mindfulness | From baseline until 6 months
  The Five Facet Mindfulness Questionnaire
Self compassion | From baseline until 6 months
  the Self Compassion Scale Short Form
Pain Catastrophizing | From baseline until 6 months
  the Pain Catastrophizing Scale
Depression and anxiety | From baseline until 6 months
  the Hospital Anxiety and Depression Scale
Well-being | From baseline until 6 months
  the WHO-5

OTHER OUTCOMES:
Attachment orientation | Baseline
  the Experiences in Close Relationships Short Version
Alexithymia | From baseline until 6 months
  the Toronto Alexithymia Scale

CONTACTS AND LOCATIONS:
Overall Officials: Maja Johannsen, PhD-fellow, MSc psychology, Principal Investigator — Unit for Psychooncology and Health Psychology, Aarhus University and Aarhus University Hospital; Robert Zachariae, Professor, MDSci., MSc, Principal Investigator — Unit for Psychooncology and Health Psychology, Aarhus University Hospital and Aarhus University
Locations (1):
- Aarhus University and Aarhus University Hospital, Aarhus, Denmark

REFERENCES:
- [Derived] Johannsen M, O'Connor M, O'Toole MS, Jensen AB, Hojris I, Zachariae R. Efficacy of Mindfulness-Based Cognitive Therapy on Late Post-Treatment Pain in Women Treated for Primary Breast Cancer: A Randomized Controlled Trial. J Clin Oncol. 2016 Oct 1;34(28):3390-9. doi: 10.1200/JCO.2015.65.0770. Epub 2016 Jun 20. PMID 27325850